CLINICAL TRIAL: NCT06834880
Title: AQT90 FLEX NTproBNP2 Test Kit - 23004 - Reference Interval Study Protocol
Brief Title: AQT90 FLEX NTproBNP2 Test Kit - 23004 - Reference Interval Study
Acronym: RI
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-087455
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy population: ADLM universal sample bank from healthy individuals are used in the study.
  Interventions: Device: No intervention; Observational study

INTERVENTIONS:
Device: No intervention; Observational study — Sample bank with Health Questionnaire

SUMMARY:
The purpose of this study is to establish the overall (age- and sex independent) at least 95th percentile upper reference limit (URL) of the NTproBNP2 Test Kit on the AQT90 FLEX analyzer.

DETAILED DESCRIPTION:
The NTproBNP2 Test is an in vitro diagnostic assay for the quantitative determination of N-terminal pro-B-type natriuretic peptide {NT-proBNP) in EDTA or lithium heparin whole blood or plasma specimens on the AQT90 FLEX analyzer in point of care/ near-patient testing and laboratory settings. It is intended for use as an aid in the diagnosis of heart failure. The test is also intended for use as an aid in the risk stratification of patients with acute coronary syndrome and heart failure.

The NTproBNP2 CAL Cartridge is an in vitro diagnostic reagent intended for the calibration adjustment of the NTproBNP2 Test on the AQT90 FLEX analyzer by establishing points of reference to estimate NT-proBNP values.

The AQT90 FLEX analyzer is an immunoassay instrument based on the quantitative determination of time-resolved fluorescence to estimate the concentrations of clinically relevant markers on whole-blood and plasma specimens to which a relevant anticoagulant has been added. It is intended for use in point of care/ near-patient testing and laboratory settings.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have given their valid consent to donate their sample in the sample bank
* Subjects must have been 18 years of age or older at the time of sample collection
* Subject must have answered yes, to being generally healthy, in the health questionnaire
* Subjects must, as a minimum, have completed questions regarding age, gender, race, and ethnicity

Exclusion Criteria:

Answered yes to any of the conditions below (Information gathered from a self-reported health questionnaire or results from blood sample tests):

* Current medications for treating cardiovascular diseases at the time of sample collection
* Current antibiotics (Indicates ongoing infections)
* Known to suffer from any of the illnesses below at the time of sample collection:

  * Disease(s) of/or affecting the cardiovascular system
  * Congestive heart failure
  * Hypertension
  * Previous history of any heart disease
  * Diabetes (Either self-reported in questionnaire or a glycosylated hemoglobin (HbA1C) in the diabetic range (above 6.4%)
  * Renal dysfunction or failure (An estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73m2.) This is to be calculated using information on age, sex and creatinine using the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation.
  * Cancer or history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 351 apparently healthy subjects in total and an approximately equal sex distribution is required for the study (i.e., approximately 50% male and 50% female population). The expected age range is from 18 and up to 90 years.
Sampling Method: Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
95th percentile of normal concentrations with 95% confidence intervals (CI) for overall samples | Baseline
  The primary endpoint of this study is to establish at least 95th percentile of normal concentrations with 95% confidence intervals (CI) for overall samples for the AQT90 FLEX NTproBNP2 Test Kit by analyzing LiHep plasma samples collected from apparently healthy subjects.

SECONDARY OUTCOMES:
95th percentile for normal concentrations separately for both males and females | Baseline
  The secondary endpoint would be to establish the 95th percentile for normal concentrations separately for both males and females with the 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiometer Turku Oy, Turku, Finland